CLINICAL TRIAL: NCT00545285
Title: Long-Term Multi-center Evaluation of E-Poly and Regenerex Cementless Acetabular Components: Clinical and Radiographic Outcomes
Brief Title: Long-Term Multi-center Evaluation of E-Poly and Regenerex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Henrik Malchau, Director of Reseach, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007P001955
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis of Hip; Traumatic Arthritis of Hip
Keywords: clinical outcomes; radiographic outcomes; total hip arthroplasty; survivorship
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Total hip Arthroplasty E-Poly™ liner in a titanium plasma sprayed RingLoc® shell
  Interventions: Procedure: Total Hip Arthroplasty
- 2 (Active Comparator): Total hip Arthroplasty ArcomXL® polyethylene liner in a titanium plasma sprayed RingLoc® shell
  Interventions: Procedure: Total Hip Arthroplasty
- 3 (Active Comparator): Total hip Arthroplasty E-Poly™ liner with Regenerex Ringloc +™ shell
  Interventions: Procedure: Total Hip Arthroplasty
- 4 (Active Comparator): Total hip Arthroplasty ArcomXL® polyethylene liner with Regenerex Ringloc +™ shell
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — Surgical implantation of specific hip replacement components for treatment of osteoarthritis

SUMMARY:
There are two distinct aims of this study:

1. This prospective study is designed to document the long-term (10-year) radiographic and clinical outcomes of a new type of highly cross-linked polyethylene liner which contains vitamin E as an anti-oxidant, (E-Poly), in a group of primary total hip arthroplasty subjects. The clinical outcome of E-Poly will be compared to a group of subjects receiving Arcom XL polyethylene.
2. This study is also designed to document the long-term (10-year) radiographic and clinical outcomes of a new cementless acetabular component having a titanium porous surface (Regenerex). The clinical outcome of this new FDA cleared device will be compared a group of subjects receiving an acetabular component having a plasma sprayed surface.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring primary total hip replacement
* Subjects with diagnosis of osteoarthritis or traumatic arthritis
* Subjects who demonstrate the ability to return for follow-up for the next 10 years

Exclusion Criteria:

* Subjects with limited life span
* Subjects with difficulty in comprehending study protocol for any reason.
* Subjects with inflammatory disease, previous infection or those requiring revision hip surgery.
* Subjects with avascular necrosis
* Subjects whose bony structures are so small that a femoral head less than 32mm in diameter must be used.
* Subjects whose bony structure deviates substantially from the general norm sufficiently to require non-standard techniques and non-standard implants. Specific examples of these are total dislocation of the hip, severe coxa vera deformity, severe forms of multiple epiphyseal dysplasia
* Subjects with complex disease entities which significantly increase the risks of the surgery such as any major platelet abnormality, hematological disorder, positive for HIV or any other major medical complication which substantially reduces longevity.
* Female subjects that are pregnant or who may suspect they are pregnant or who plan to become pregnant while participating in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-11; Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Survivorship: length of time implant remains without revision | Evaluated at 1,3,5,7 ,10th year over 10 years
Complications and Adverse Events | Evaluated at 1,3,5,7 ,10th year over 10 years
Incidence of radiolucencies (acetabular component) | Evaluated at 1,3,5,7 ,10th year over 10 years
Patient administered Outcome Survey scores | Evaluated at 1,3,5,7 ,10th year over 10 years
Polyethylene wear rates from AP radiographs | Evaluated at 1,3,5,7 ,10th year over 10 years

SECONDARY OUTCOMES:
Survivorship in subcategories of infection, aseptic loosening and other | 1,3,5,7,10 yr over 10 years
Subcategories of the outcome scores regarding pain, patient satisfaction, function,general quality of life. | 1,3,5,7,10 yr over 10 years
Other outcomes that may be relevant. | 1,3,5,7,10 yr over 10 years
Retrieval analysis | 1,3,5,7,10 yr over 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Malchau, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sillesen NH, Greene ME, Nebergall AK, Huddleston JI, Emerson R, Gebuhr P, Troelsen A, Malchau H. 3-year follow-up of a long-term registry-based multicentre study on vitamin E diffused polyethylene in total hip replacement. Hip Int. 2016 Jan-Feb;26(1):97-103. doi: 10.5301/hipint.5000297. Epub 2015 Dec 11. PMID 26692248